CLINICAL TRIAL: NCT06599814
Title: Comparative Evaluation of the Clinical Outcome of Direct Pulp Capping Treatment Using Bioactive Materials With Diode Laser in Permanent Molars: a Randomized Clinical Trial
Brief Title: Comparative Evaluation of the Clinical Outcome of Direct Pulp Capping Treatment in Permanent Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hisham Mahmoud Hamdy Abada, lecturer of Endodontics, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-245
Record Dates: First submitted 2024-06-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vital Pulp Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RetroMTA Conventional group (Active Comparator): After controlling the bleeding, RetroMTA is mixed with the supplied liquid at a W/P ratio of 3 drops per 0.3 g. After 150 seconds, selective etching, application of adhesive material and application of resin composite restorations will occur according to the manufacturer's instructions.
  Interventions: Procedure: vital pulp therapy
- TheraCal Conventional group (Active Comparator): Subsequent to controlling the bleeding, using a needle-tip syringe, gently apply TheraCal LC resin-modified calcium silicate (Bisco Inc., Schamburg, IL, USA) light-hardening paste to the exposed portion of the pulp in accordance with the manufacturer's recommendations for thickness (1 mm) and curing time (20 Seconds).
  Interventions: Procedure: vital pulp therapy
- RetroMTA laser group (Active Comparator): Consequent to controlling the bleeding, Diode laser is focused to the exposure sites before the placement of pulp capping materials. The hemostasis is obtained by the diode 808-nm, laser-assisted procedure (Picasso-AMD, USA) using 1.5 W, continuous wave, fiber diameter of 400 μm, non-initiated and in contact mode, Decontamination of the cavity is performed by 1 W, continuous wave, fiber diameter of 400 μm, non-initiated and in contact mode, tip angle set at 90°, an area with 2-mm diameter per second, power density 31.83 W/cm2, energy density 31.83 J/cm2 per second (28), and circular movement (23). The use of diode laser will be used for 1 to 3 Application of RetroMTA are occurred as RetroMTA Conventional group.
  Interventions: Procedure: vital pulp therapy
- TheraCal laser group (Active Comparator): Consequent to controlling the bleeding, Diode laser is focused to the exposure sites before the placement of pulp capping materials. The hemostasis is obtained by the diode 808-nm, laser-assisted procedure (Picasso-AMD, USA) using 1.5 W, continuous wave, fiber diameter of 400 μm, non-initiated and in contact mode, Decontamination of the cavity is performed by 1 W, continuous wave, fiber diameter of 400 μm, non-initiated and in contact mode, tip angle set at 90°, an area with 2-mm diameter per second, power density 31.83 W/cm2, energy density 31.83 J/cm2 per second (28), and circular movement (23). The use of diode laser will be used for 1 to 3 Application of TheraCal are occurred as TheraCal Conventional group.
  Interventions: Procedure: vital pulp therapy

INTERVENTIONS:
Procedure: vital pulp therapy — vital pulp therapy using two bioactive materials TheraCal and RetroMTA as direct pulp caping materials conventionally and test using Diode laser before application of these materials

SUMMARY:
This clinical trial will be performed during June 2024 and December 2024. The study is conducted following the Declaration of Helsinki Ethical principles for medical research involving human subjects after being independently reviewed and approved by the Institution's Ethical Committee and is designed in accordance with CONSORT 2010.

Selected patients who are between 19 and 40 years of age had undergone conservative treatment for deep caries management in their permanent teeth in the restorative and endodontic departments, faculty of dentistry, Kafrelsheikh university. The patients are then assigned randomly into four different groups for this randomized clinical study. The decision for direct pulp capping will be made after informing the patients about all the pulp capping procedures that are suggested. Furthermore, any possible complications, postoperative discomfort, or failure of the treatment will be discussed with the patient. All included patients signed a written informed consent before enrollment

DETAILED DESCRIPTION:
A total of 120 posterior teeth from 60 patients are randomly divided into 4 groups according to the type of treatment; RetroMTA Conventional group, TheraCal Conventional group, RetroMTA laser group, and TheraCal laser group (n = 30).

A checklist is created for each patient following their selection and completion of the consent form. periapical radiography is carried out and cold/heat tests, to confirm the vitality of the teeth. Mouth rinsing is done with 0.2% chlorhexidine oral rinse for 1 minute. All of the patients' teeth are treated by the same dentist. In all groups, if the bleeding persisted for longer than three minutes following pulp exposure would be eliminated from the research.

Clinical procedures Following local anesthetic, the teeth are suitably isolated under a rubber dam and the caries is removed using the appropriate hand and rotating equipment. There will have been tooth cleaning and bleeding control using cotton pellets lightly moistened with sterile saline applied to the exposed site. Patients are randomly divided into two techniques; a conventional technique that acts as a control group in which laser is not used, and a laser-assisted technique in which Diode laser is applied before application of pulp capping materials. The patients are allocated into one of the following groups; RetroMTA Conventional group, TheraCal Conventional group, RetroMTA laser group, and TheraCal laser group.

Conventional Technique (control group) RetroMTA Conventional group (n = 30). After controlling the bleeding, RetroMTA is mixed with the supplied liquid at a W/P ratio of 3 drops per 0.3 g. After 150 seconds, selective etching, application of adhesive material and application of resin composite restorations will occur according to the manufacturer's instructions.

TheraCal Conventional group (n = 30). Subsequent to controlling the bleeding, using a needle-tip syringe, gently apply TheraCal LC resin-modified calcium silicate (Bisco Inc., Schamburg, IL, USA) light-hardening paste to the exposed portion of the pulp in accordance with the manufacturer's recommendations for thickness (1 mm) and curing time (20 Seconds).

Laser-assisted technique Consequent to controlling the bleeding, Diode laser is focused to the exposure sites before the placement of pulp capping materials. The protective goggles for the patient, operator, and assistant are checked. The hemostasis is obtained by the diode 808-nm, laser-assisted procedure (Picasso-AMD, USA) using 1.5 W, continuous wave, fiber diameter of 400 μm, non-initiated and in contact mode, tip angle set at 90°, beam divergence 16°, 2 s per an area with 1-mm diameter, power density 190.98 W/cm2, energy density 381.97 J/cm2, and vertical and horizontal scanning movement on the exposure site. Decontamination of the cavity is performed by 1 W, continuous wave, fiber diameter of 400 μm, non-initiated and in contact mode, tip angle set at 90°, an area with 2-mm diameter per second, power density 31.83 W/cm2, energy density 31.83 J/cm2 per second, and circular movement. The use of diode laser will be used for 1 to 3 seconds. Following to laser application, the pulp capping materials either RetroMTA or TheraCal are placed over the exposure site according to the randomization protocol.

TheraCal laser group (n = 30). Application of TheraCal are occurred as TheraCal Conventional group. RetroMTA laser group (n = 30). Application of RetroMTA are occurred as RetroMTA Conventional group. Restorative procedures The cavities are permanently restored at the same session using universal Adhesive in selective etch technique for enamel margins and self-etch for cavities dentine following a layer of flowable and then nanohybrid composite.

Follow-Up and Evaluation of the Success At each recall examination (1, 3, and 6 months), the information obtained from clinical and radiographic examinations is recorded in a special form. Clinical assessments are performed by applying ice on the buccal side, percussion test to forecast the periradicular involvement of the tooth, and palpation test to forecast the extent of periradicular bone involvement. In addition, follow up of the postoperative pain will be occurred. The clinical failure criteria included the loss of vitality, spontaneous pain, prolonged reactions to thermal stimuli, and tenderness to percussion.

Radiographic assessments are performed by a calibrated endodontist who is also blind to the type of treatment groups. Every digital radiograph is examined for dentin formation, periapical and furcal radiolucency, expansion of the periodontal ligament space, and any pulpal calcifications. After that, every radiograph is scanned and uploaded to the computer for digital analysis. Measurements on the digitized radiographs are performed in the first, third, and sixth months. The increase in dentin thickness is thus measured using Image J program (Microsoft Corp®, Washington, Redmond, USA). The statistical analyses based on the repeated measurements ANOVA are conducted for selected data sets.

ELIGIBILITY:
Inclusion Criteria:

* In all patients, the pulp had been exposed because of caries removal. Data collection included clinical pulp capping respecting the following criteria.

Exclusion Criteria:

1. Individuals who are 19 to 40 years old.
2. Permanent teeth that have not been repaired and have extensive caries on their occlusal and proximal surfaces, extending more than two-thirds of the dentin near the pulp.
3. Vital teeth; asymptomatic teeth (not sensitive to pressure, percussion, or palpation, and no spontaneous pain); sinus tract devoid of swelling and abscess; abnormal mobility absent; no history of spontaneous pain; mild, dull, and tolerable pain associated with eating and drinking cold drinks.
4. Ethyl chloride cold tests, gutta-percha heat testing, palpation, percussion, and the lack of radiological symptoms in periapical radiographs are used to assess the life of the teeth prior to treatment. After the stimulus is removed, pain from a pulp test that is triggered by either heat or cold should subside.
5. In periapical radiography, none of the following conditions should be present: normal lamina dura and periodontal ligaments, no internal or external root resorption, and no radiolucency in the furcation area or periapical region.
6. The exposed area's diameter ranges from 0.5 to 1 mm.
7. Participants' acceptance of the research program.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | (1, 3, and 6 months
  The postoperative pain was assessed on the numeric rating scale (NRS-11) 1,3 and 6 months after intervention. The examiner asked the patient to quantify his/her maximum pain intensity within the last 24 hours on a scale of 0 to 10. The following anchors were used to describe the rating scale: 0 = no pain/pain-free and 10 = worst pain imaginable.
Radiographic assessments | (1, 3, and 6 months
  The digital periapical radiographs were captured using a paralleling technique with Rinn film holders to allow standardization. Each root was examined for the presence, absence, and change (increase/decrease) in size of any PA radiolucency. A PA lesion or PDL gap expansion was referred to as a PA radiolucency. Less than double the equal healthy PDL space of the neighboring healthy tooth was considered a widening of the PDL space. A PA lesion was identified as radiolucency connected to the root's radiographic apex, greater than double the PDL space's breadth

CONTACTS AND LOCATIONS:
Locations (1):
- kafrelsheikh University, Kafr ash Shaykh, Kafr El-Shaikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided